CLINICAL TRIAL: NCT03888833
Title: Risk Factors of Bleeding in Patients Undergoing Peripheral Veno Arterial Extra Corporeal Membrane Oxygenation
Brief Title: Risk Factors of Bleeding Under Veno Arterial Membrane Oxygenation
Acronym: ECMO bleeding
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: ELLOUZE 2019
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Extracorporeal Membrane Oxygenation; Bleeding; Complication
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Veno arterial extracorporeal membrane oxygenation
  Interventions: Device: ECMO

INTERVENTIONS:
Device: ECMO — ECMO installation

SUMMARY:
Veno arterial extracorporeal membrane oxygenation (VA ECMO) is used, for cardiogenic shock, refractory cardiac arrest and post cardiotomy cardiac failure. Bleeding is frequent complications during VA ECMO and is associated with increased mortality. The aim of our study was to identify early factors associated with major bleeding in patients supported by VA ECMO

ELIGIBILITY:
Inclusion Criteria: Patients over 18 years treated by peripheral veno arterial membrane oxygenation

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veno arterial extracorporeal membrane oxygenation
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Rate of major hemorrhagic episodes defined as follows: loss of over 2g dl-1 of hemoglobin in 24 h, bleeding rate over 20 ml kg-1 day-1 or blood transfusion over 10 ml kg-1 day-1 | Through study completion, an average of 10 years
  Our main objective was to evaluate risk factors independently associated with major hemorrhagic episode. We collected patient characteristics at the start of VA ECMO: age, gender, anthropometric information, medical history and chronic treatments. We also calculated SOFA and APACHE II scores on the day of VA ECMO implementation. We noted the indication for VA ECMO, any pre-cannulation treatments (fibrinolysis, aspirin, heparin), where VA ECMO was inserted and whether or not an intra-aortic balloon pump was present. With regard to various complications, we collected the quantity of delivered blood products , the site of bleeding initial temperature. The biological data were collected at initiation of VA ECMO.

SECONDARY OUTCOMES:
Rate of mortality | 30 day
Duration of life support | Through study completion, an average of 10 years
Length of stay | Through study completion, an average of 10 years
Ischemic and thrombotic complications | Through study completion, an average of 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Ellouze O, Abbad X, Constandache T, Missaoui A, Berthoud V, Daily T, Aho S, Bouchot O, Bouhemad B, Guinot PG. Risk Factors of Bleeding in Patients Undergoing Venoarterial Extracorporeal Membrane Oxygenation. Ann Thorac Surg. 2021 Feb;111(2):623-628. doi: 10.1016/j.athoracsur.2020.02.012. Epub 2020 Mar 12. PMID 32171730